CLINICAL TRIAL: NCT00799305
Title: Correlation of Airflow Limitation and Other Respiratory Characteristics With Radiologic Changes of Lung Structure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Marinella Beckerman, Internal Medicine Dept. Hillel Yaffe Medical Center
Other Study IDs: 0046-08-HYMC
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COPD patients

SUMMARY:
The aim of the study is to assess the correlation between airflow limitation, perception of dyspnea and functional capacity with anatomic changes in pulmonary structure as seen on High Resolution CT in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Able to perform pulmonary function testing

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD attending pulmonary clinic in the internal disease department at the Hillel Yaffe Medical Center
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-01

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel